CLINICAL TRIAL: NCT06737965
Title: Cardiovascular Immaturity in Extremely Low Gestational Age Newborns: a Fundamental Prospective Study
Acronym: ELGAN AMINES
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM U1046 Physiologie et médecine expérimentale du coeur et des muscles (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0118; AO Tremplin (Other Grant/Funding Number: CHU de Montpellier)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-10

CONDITIONS: ELGAN (22-28SA); Extremely Low Gestational Age Newborns; Cardiovascular Immaturity
Keywords: Cardiovascular immaturity in extremely premature infants; vasoactive agent; vascular reactivity; cardiac adrenergic receptor; cardiac architecture; vascular response; Extremely low gestational age newborns; cardio-circulatory insufficiency; myocardial contraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Extremely low gestational age foetuses: Material (cord blood/myocardial tissu/ vascular segment) from foetuses resulting from medical abortion before 28 weeks of gestation (and after 22 weeks of gestation)
  Interventions: Other: Medical abortion; Other: Foetopathology exam; Other: Outcomes mesurement
- Control group : foetuses ≥ 34 weeks of gestation: Material (cord blood/myocardial tissu/ vascular segment) from foetuses resulting from medical abortion after or during 34 weeks of gestation
  Interventions: Other: Medical abortion; Other: Foetopathology exam; Other: Outcomes mesurement

INTERVENTIONS:
Other: Medical abortion — Medical abortion performed according to standard practice with cord blood sample (1 to 10ml) collected on EDTA tube before injection of foeto toxic agent.
  EDTA tube transfered to laboratory on ambient temperature. Blood sample will be centrifuged to isolate the extracellular vesicles once in the laboratory.
  Other Names: Cord blood sample / Blood analyse
Other: Foetopathology exam — Foetopathology exam is performed according to standard practice on the day after abortion (H12 to H48 from foetus death).
  Investigator will recover 2 horizontal slices (in line with the heart) between 3 and 5 mm thick, including the right and left ventricles put them in a cold physiological saline solution, and transfer them rapidly to the laboratory.
  Investigator will also recover segments of the descending aorta (approximately 2cm, between the ductus arteriosus and the celiac trunk) and the left renal artery. The isolated segments will be separated from the fat and connective tissue by the foetopathology team and put in a cold physiological saline solution.
  Other Names: Sampling of myocardial tissue and vascular segments
Other: Outcomes mesurement — * From the myocardial samples, 10 µm thick sections will be prepared and slides will be incubated with antibodies directed against proteins of interest (adrenergic receptors, protein kinase A, ryanodine receptor, PDE3, troponin). After washing, fluorescent secondary antibodies will be used and slides will be observed under a fluorescence microscope. Rest of the cardiac tissue will be frozen in liquid nitrogen in order to perform Western blots.
  * Vessel samples will be put in a myograph to study contractile function. Concentration-response curves will be constructed by cumulative application of noradrenaline or U46619. For the study of endothelial function, arteries with and without functional endothelium will be pre-contracted to 80% of maximal contraction with U46619. When contraction reaches a plate, cumulative addition of different vasodilating agents will be performed. The vessels will also be cannulated on an arteriograph to assess dilation in response to flow and myogenic tone.

SUMMARY:
Birth is a major turning point in the life of the newborn, as it moves from intrauterine life to extrauterine life. This sudden transition forces the newborn to adapt quickly. Oxygenation, which was only provided by the placenta during uterine life, will have to be provided by the lungs, which will open when the newborn cries for the first time. This phenomenon will change the way blood reaches the lungs and will require the newborn's heart to work harder. In addition, the cardiac workload will also increase due to the clamping of the umbilical cord, which will force the heart to pump through more resistant blood vessels.

This transition, generally well tolerated in newborns at term, can be much more complicated in premature newborns, particularly in extremely low gestational age newborns (e.g. ELGAN, born before 28 weeks of amenorrhoea). There are several causes of this difficult adaptation on the cardiovascular system: poor heart function, difficulty in revascularizing lungs due to the physiological characteristics of premature newborns (high pulmonary vascular resistance, persistence of the ductus arteriosus), and a tone of the blood vessel muscles that is probably immature. In addition, respiratory failure is often associated with pulmonary immaturity.

The consequences of a difficult adaptation to extrauterine life, combined with cardiovascular failure, will be poor organ perfusion, whose brain. Moreover, ELGANs have immature regulation of their brain vascularisation. Variations in the vascularisation of the brain (in the event of cardiovascular failure) may be responsible for irreversible lesions with intraventricular hemorrhage. Ultimately, these bleedings carry a high risk of mortality or severe disability in premature infants.

Several hypotheses have been put forward as to the causes of this poor adaptation to extrauterine life, but there are few recommendations on adapted medical management. Cardiac ultrasound and the use of drugs to support the heart and blood vessels have been suggested. However, a large number of ELGANs will develop complications that investigators cannot predict or intervene in time. In addition, studies on the drugs used have not been carried out on ELGANs, which limits the conclusions investigators can draw.

These factors encourage us to improve our fundamental knowledge of the cardiovascular system in the ELGANs. The aim is to identify the most effective clinical tools and treatments for assessing and treating neonatal cardiovascular failure at an early stage, before complications appear. Investigators aim to compare the architecture and composition of the heart, blood vessels, and blood of fetuses under 28 weeks of amenorrhea gestation with those of fetuses over or equal to 34 weeks of amenorrhea gestation.

For this research, investigators need tissues (heart muscle, blood, and vessels) from fetuses of different ages. These tissues are usually already taken during the foetopathology examination to try to provide a medical explanation of the medical abortion. There will be no change to the foetopathology examination carried out on the foetus, with the exception that some of the tissue taken will have additional analyses carried out in our INSERM laboratory attached to the Montpellier University Hospital.

Population resulting from medical abortion is motivated by the ethical impossibility of taking such invasive samples from live newborns. The non-use of animals is justified by the difficulty of extrapolating results to humans. The indication for abortion and its performance will be carried out by current practice. Participants will be offered and explained the study during the pre abortion visit.

This research does not alter the patient's care. No additional examination or consultation is required. No personal benefit is expected from the study, but it will enable us to gain a better understanding of ELGAN's hemodynamics and to consider future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

For the pregnant women:

* Over 18 years old.
* Speaks and understands French.
* Medical abortion requested by the participant, scheduled and validated by the CPDPN of the Montpellier University Hospital.
* Participant's agreement to use for research purposes the biological tissues from the systematic foetopathological examination.

For fetuses:

* Interest group: Fœtus ≥ 22 WA and <28 WA
* Control group: Fœtus ≥ 34 WA

Exclusion Criteria:

For the pregnant women :

* Injection of betamethasone or maternal use of dexamethasone in the month before foeticide
* Known family genetic mutation that may be linked with cardiomyopathy
* Failure to obtain consent (adults, unemancipated minors, persons unable to give consent)
* Not affiliated to a social security
* Persons under legal protection
* Person taking part in another research study with an exclusion period still in progress.

For fetuses:

* Fetus from unplanned in-utero death
* Significant cardiac malformation suspected antenatally (excluding atrial septal defect ostium secundum and isolated muscular ventricular septal defect).
* Suspected abnormality of myocardial tissue
* Biological tissue sampling more than 48 hours after fœticide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pregnant woman who will receive a medical abortion at Montpellier Hospital and who present eligibility criteria for her and her foetus will be invited to participate to the study
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the quantity of beta adrenergic receptor linked to myocardial contraction according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of beta-adrenergic receptor
  - ß-adrenergic receptor levels: ß-adrenergic expression / GAPDH (Glyceraldehyde-3-phosphate dehydrogenase) expression. Expressed as a percentage
Comparison of the quantity of phosphodiesterase 3 linked to myocardial contraction according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of the quantity of phosphodiesterase 3 (PDE3) :
  - Phosphodiesterase 3 levels: PDE3 expression / Glyceraldehyde-3-phosphate dehydrogenase (GAPDH) expression. Expressed as a percentage

SECONDARY OUTCOMES:
Comparison of the quantity of cyclic AMP linked to myocardial contraction according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of quantity of cyclic AMP (adenosine monophosphate) levels. Expressed in pm/mL.
Comparison of the quantity of protein kinase A linked to myocardial contraction according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of the quantity of protein kinase A levels. Expressed in U/mL.
Comparison of the quantity of type 2 ryanodine receptor linked to myocardial contraction according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of the type 2 Ryanodine receptor levels (RyR2): RyR 2 expression / Glyceraldehyde-3-phosphate dehydrogenase (GAPDH) expression. Expressed as a percentage
Comparison of the quantity of troponin linked to myocardial contraction according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of the troponin levels (troponin I, C and T): Troponin expression / Glyceraldehyde-3-phosphate dehydrogenase (GAPDH) expression. Expressed as a percentage
Comparison of the vascular response of smooth muscle according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of vascular response on the aorta and renal artery: smooth muscle contractile function. Expressed in mN/mm
Comparison of the vascular response of myogenic tone according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of vascular response on the aorta and renal artery: myogenic tone. Expressed in um
Comparison of the vascular response of endothelial function according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of vascular response on the aorta and renal artery: endothelial function. Expressed as percentage
Comparison of the myocardial architecture according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of myocardial architecture.
Comparison of the vasoactive agents level in blood according to the term of foetal death | Within 48 hours of the abortion
  Comparison between the two groups of vasoactive agents level by measuring the level of extracellular vesicles in cord blood. Expressed as a percentage.
Comparison of the vascular alpha adrenergic receptor levels according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of alpha adrenergic receptor levels on vascular segment (percentage)
Comparison of the cytosolic and mitochondrial oxidative stress according to the term of foetal death | After foetopathology exam within 48 hours of the abortion
  Comparison between the two groups of cytosolic and mitochondrial oxidative stress (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Osborn DA, Paradisis M, Evans N. The effect of inotropes on morbidity and mortality in preterm infants with low systemic or organ blood flow. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD005090. doi: 10.1002/14651858.CD005090.pub2. PMID 17253539
- [Background] Subhedar NV, Shaw NJ. Dopamine versus dobutamine for hypotensive preterm infants. Cochrane Database Syst Rev. 2003;(3):CD001242. doi: 10.1002/14651858.CD001242. PMID 12917901
- [Background] Raschetti R, Torchin H, Marchand-Martin L, Gascoin G, Cambonie G, Brissaud O, Roze JC, Storme L, Ancel PY, Mekontso-Dessap A, Durrmeyer X. In-hospital Outcomes and Early Hemodynamic Management According to Echocardiography Use in Hypotensive Preterm Infants: A National Propensity-Matched Cohort Study. Front Cardiovasc Med. 2022 Jul 14;9:852666. doi: 10.3389/fcvm.2022.852666. eCollection 2022. PMID 35911541
- [Background] Roze JC, Cambonie G, Marchand-Martin L, Gournay V, Durrmeyer X, Durox M, Storme L, Porcher R, Ancel PY; Hemodynamic EPIPAGE 2 Study Group. Association Between Early Screening for Patent Ductus Arteriosus and In-Hospital Mortality Among Extremely Preterm Infants. JAMA. 2015 Jun 23-30;313(24):2441-8. doi: 10.1001/jama.2015.6734. PMID 26103028
- [Background] Mertens L, Seri I, Marek J, Arlettaz R, Barker P, McNamara P, Moon-Grady AJ, Coon PD, Noori S, Simpson J, Lai WW; Writing Group of the American Society of Echocardiography; European Association of Echocardiography; Association for European Pediatric Cardiologists. Targeted Neonatal Echocardiography in the Neonatal Intensive Care Unit: practice guidelines and recommendations for training. Writing Group of the American Society of Echocardiography (ASE) in collaboration with the European Association of Echocardiography (EAE) and the Association for European Pediatric Cardiologists (AEPC). J Am Soc Echocardiogr. 2011 Oct;24(10):1057-78. doi: 10.1016/j.echo.2011.07.014. No abstract available. PMID 21933743
- [Background] de Waal K, Evans N. Hemodynamics in preterm infants with late-onset sepsis. J Pediatr. 2010 Jun;156(6):918-922.e1. doi: 10.1016/j.jpeds.2009.12.026. Epub 2010 Mar 16. PMID 20236658
- [Background] Batton B, Li L, Newman NS, Das A, Watterberg KL, Yoder BA, Faix RG, Laughon MM, Stoll BJ, Van Meurs KP, Carlo WA, Poindexter BB, Bell EF, Sanchez PJ, Ehrenkranz RA, Goldberg RN, Laptook AR, Kennedy KA, Frantz ID 3rd, Shankaran S, Schibler K, Higgins RD, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health & Human Development Neonatal Research Network. Use of antihypotensive therapies in extremely preterm infants. Pediatrics. 2013 Jun;131(6):e1865-73. doi: 10.1542/peds.2012-2779. Epub 2013 May 6. PMID 23650301
- [Background] Giesinger RE, Rios DR, Chatmethakul T, Bischoff AR, Sandgren JA, Cunningham A, Beauchene M, Stanford AH, Klein JM, Ten Eyck P, McNamara PJ. Impact of Early Hemodynamic Screening on Extremely Preterm Outcomes in a High-Performance Center. Am J Respir Crit Care Med. 2023 Aug 1;208(3):290-300. doi: 10.1164/rccm.202212-2291OC. PMID 37209133
- [Background] Aldana-Aguirre JC, Deshpande P, Jain A, Weisz DE. Physiology of Low Blood Pressure During the First Day After Birth Among Extremely Preterm Neonates. J Pediatr. 2021 Sep;236:40-46.e3. doi: 10.1016/j.jpeds.2021.05.026. Epub 2021 May 18. PMID 34019882
- [Background] Sakurai K, Takeba Y, Osada Y, Mizuno M, Tsuzuki Y, Aso K, Kida K, Ohta Y, Ootaki M, Iiri T, Hokuto I, Shimizu N, Matsumoto N. Antenatal Glucocorticoid Administration Promotes Cardiac Structure and Energy Metabolism Maturation in Preterm Fetuses. Int J Mol Sci. 2022 Sep 5;23(17):10186. doi: 10.3390/ijms231710186. PMID 36077580
- [Background] Osborn DA, Evans N, Kluckow M. Left ventricular contractility in extremely premature infants in the first day and response to inotropes. Pediatr Res. 2007 Mar;61(3):335-40. doi: 10.1203/pdr.0b013e318030d1e1. PMID 17314693
- [Background] Seidler AL, Gyte GML, Rabe H, Diaz-Rossello JL, Duley L, Aziz K, Testoni Costa-Nobre D, Davis PG, Schmolzer GM, Ovelman C, Askie LM, Soll R; INTERNATIONAL LIAISON COMMITTEE ON RESUSCITATION NEONATAL LIFE SUPPORT TASK FORCE. Umbilical Cord Management for Newborns <34 Weeks' Gestation: A Meta-analysis. Pediatrics. 2021 Mar;147(3):e20200576. doi: 10.1542/peds.2020-0576. PMID 33632931
- [Background] Kluckow M, Evans N. Low superior vena cava flow and intraventricular haemorrhage in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2000 May;82(3):F188-94. doi: 10.1136/fn.82.3.f188. PMID 10794784
- [Background] Hunt RW, Evans N, Rieger I, Kluckow M. Low superior vena cava flow and neurodevelopment at 3 years in very preterm infants. J Pediatr. 2004 Nov;145(5):588-92. doi: 10.1016/j.jpeds.2004.06.056. PMID 15520755
- [Background] Treluyer L, Chevallier M, Jarreau PH, Baud O, Benhammou V, Gire C, Marchand-Martin L, Marret S, Pierrat V, Ancel PY, Torchin H. Intraventricular Hemorrhage in Very Preterm Children: Mortality and Neurodevelopment at Age 5. Pediatrics. 2023 Apr 1;151(4):e2022059138. doi: 10.1542/peds.2022-059138. PMID 36919442
- [Background] Papile LA, Burstein J, Burstein R, Koffler H. Incidence and evolution of subependymal and intraventricular hemorrhage: a study of infants with birth weights less than 1,500 gm. J Pediatr. 1978 Apr;92(4):529-34. doi: 10.1016/s0022-3476(78)80282-0. PMID 305471
- [Background] Boylan GB, Young K, Panerai RB, Rennie JM, Evans DH. Dynamic cerebral autoregulation in sick newborn infants. Pediatr Res. 2000 Jul;48(1):12-7. doi: 10.1203/00006450-200007000-00005. PMID 10879794
- [Background] Kozlik R, Kramer HH, Wicht H, Krian A, Ostermeyer J, Reinhardt D. Myocardial beta-adrenoceptor density and the distribution of beta 1- and beta 2-adrenoceptor subpopulations in children with congenital heart disease. Eur J Pediatr. 1991 Apr;150(6):388-94. doi: 10.1007/BF02093715. PMID 1645667
- [Background] Paradisis M, Osborn DA. Adrenaline for prevention of morbidity and mortality in preterm infants with cardiovascular compromise. Cochrane Database Syst Rev. 2004;2004(1):CD003958. doi: 10.1002/14651858.CD003958.pub2. PMID 14974048
- [Background] Ibrahim H, Sinha IP, Subhedar NV. Corticosteroids for treating hypotension in preterm infants. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD003662. doi: 10.1002/14651858.CD003662.pub4. PMID 22161379
- [Background] Cambonie G, Clyman RI, Roze JC. Management of persistent ductus arteriosus in very premature neonates. Results of the French TRIOCAPI trial, perspectives for clinicians, and subsequent studies on this topic. Arch Pediatr. 2021 Oct;28(7):501-503. doi: 10.1016/j.arcped.2021.07.002. Epub 2021 Sep 9. No abstract available. PMID 34511277
- [Background] Mitra S, de Boode WP, Weisz DE, Shah PS. Interventions for patent ductus arteriosus (PDA) in preterm infants: an overview of Cochrane Systematic Reviews. Cochrane Database Syst Rev. 2023 Apr 11;4(4):CD013588. doi: 10.1002/14651858.CD013588.pub2. PMID 37039501
- [Background] Evans N. Assessment and support of the preterm circulation. Early Hum Dev. 2006 Dec;82(12):803-10. doi: 10.1016/j.earlhumdev.2006.09.020. Epub 2006 Oct 31. PMID 17079097
- [Background] Paradisis M, Evans N, Kluckow M, Osborn D. Randomized trial of milrinone versus placebo for prevention of low systemic blood flow in very preterm infants. J Pediatr. 2009 Feb;154(2):189-95. doi: 10.1016/j.jpeds.2008.07.059. Epub 2008 Sep 25. PMID 18822428
- [Background] Noori S, Seri I. Hemodynamic antecedents of peri/intraventricular hemorrhage in very preterm neonates. Semin Fetal Neonatal Med. 2015 Aug;20(4):232-7. doi: 10.1016/j.siny.2015.02.004. Epub 2015 Mar 27. PMID 25818879